CLINICAL TRIAL: NCT02126072
Title: The Effects of Ethanol on Gut Wall Integrity as Measured by I-FABP and LBP
Brief Title: Effects of Ethanol on Gut Wall Integrity
Acronym: E-GUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, JBF Hulscher, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2011/262
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Alcohol Consumption
Keywords: Ethanol; Alcohol; Consumption; Gut wall integrity; Endotoxemia
MeSH Terms: conditions — Alcohol Drinking; Endotoxemia | interventions — Ethanol; Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol (Experimental): The study is a randomized single blinded trial in cross over design. Subjects are randomized to drink alcohol in one session and water in another session.
  Interventions: Dietary Supplement: Alcohol
- Water (Active Comparator): Water in the same volume as the volunteer would have to drink in wine according to the protocol.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Alcohol — They consume 1gram of alcohol per kilogram of bodyweight in wine (12%)
  Arms: Alcohol
Dietary Supplement: Water — Volunteers consume the same volume of water as the would in wine according toe the protocol.
  Arms: Water

SUMMARY:
Objective: To determine the immediate effects of oral alcohol consumption in healthy volunteers on gut wall integrity as measured by I-FABP and LBP.

Study design: Randomized, single blinded cross over study.

Study population: 15 healthy adult male human volunteers will be included in this study.

Intervention: the consumption of alcoholic beverages (1 g/kg ethanol) of wine (12%) compared to the consumption of water.

Main study parameters/endpoints: The aim of this study is to determine the immediate effects of oral alcohol consumption in healthy volunteers on gut wall integrity as measured by I-FABP and LBP.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects consume 1g of alcohol per kg bodyweight. One blood sample of 14 ml followed by 6 samples of 8 ml will be drawn between 16.45 hours and 19:00 hours the day after. The first 6 observations take place in a single visit followed by one observation in short visit the next day. It is unlikely that subjects will experience any physical or psychological discomfort from the withdrawal of a total of 62 ml of blood in 24 hours or the consumption of the amounts alcohol or water mentioned above. The same protocol will be repeated one week after the first visit in which the alcohol group and water group are crossed over.

DETAILED DESCRIPTION:
A common finding in trauma patients admitted to the ER with serious injuries is the presence of alcohol abuse. Alcohol is involved in up to 40% of deaths from motor vehicle crashes, 60% of deaths from intentional injuries, and 50% of hospital admissions for injuries.

Chronic alcohol consumption leads to a decrease in gut wall integrity in actively drinking alcoholics and patients with alcohol induced liver disease. Animal studies show that the mucosal damage caused by alcohol consumption increases the permeability of the gut to macromolecules. This facilitates the translocation of endotoxin and other bacterial toxins from the gut lumen to the portal circulation. In addition to increased endotoxemia other studies show that the initial event in response to alcohol is an increased influx of leukocytes leading to an enhanced release of noxious mediators, such as reactive oxygen species, leukotrienes and histamine by mast cells. Alcohol consumption thus leads to a decrease in gut wall integrity with increased endotoxemia and as a result induces an inflammatory response. Data on the effects of acute alcohol consumption on gut wall integrity in non-alcoholics is still scarce.

In patients exposed to severe trauma, loss of gut wall integrity has been implicated as an important contributor to the development of excessive inflammation [6]. Intestinal mucosal damage develops early after trauma leading to loss of gut wall integrity and resulting in translocation of luminal bacteria and toxins into the gut wall. This has been associated with the development of an inflammatory response. This excessive inflammation can in turn lead to the systemic inflammatory response syndrome (SIRS) which can ultimately lead to multiple organ failure (MOF) and death. Up to 20% of the deaths in trauma patients are due to the consequences of SIRS and MOF.

When assessing the effects of alcohol and severe trauma on gut wall integrity combined with the fact that the two co-exist frequently one can hypothesize that the outcome for trauma patients under the influence of alcohol is detrimental. Literature regarding this issue is unequivocal, consisting only of relatively small retrospective series.

Population (base) 15 healthy adult male human volunteers will be included in this study

Inclusion criteria

* male volunteers
* age between 18 and 60 years
* written informed consent

Exclusion criteria

* medical history of alcohol abuse
* use of any medication
* medical history of bowel disease

Volunteers will confirm meeting the inclusion criteria by signing the informed consent.

Sample size calculation As there is currently no data available on the effect of alcohol on gut wall integrity as measured by FABP the investigators will conduct a pilot study. The chosen population size of 15 volunteers is based upon financial and organisational benefits.

Investigational product/treatment Subjects will consume either 1g/kg of wine (12%) or 600 ml of water within 45 minutes.

METHODS Main study parameter/endpoint Primary Objective: The aim of this study is to determine the immediate effects of oral alcohol consumption in healthy volunteers on gut wall integrity as measured by I-FABP and LBP.

The gut wall integrity will be assessed using I-FABP as a measure of the integrity of the enterocyte. Lipopolysaccharide binding protein (LBP), a protein that binds LPS, will serve as a measure of endotoxemia. Furthermore, the effect of alcohol on gut wall integrity markers per se is assessed by artificially adding alcohol to blood and comparing it to non-alcoholised blood.

The following 'patient' characteristics are acquired to assess their possible effect on FABP/LBP levels and to correct for any variance that is witnessed: age, weight, length, body temperature and race.

Study procedures After informed consent fifteen healthy adult male volunteers, aged 18-60, will participate in the study. They will be randomized into two groups: one will consume alcohol, the other will consume water (see below). One week later, the groups will switch Volunteers with a medical history of alcohol abuse or bowel disease or subjects using any medication will be excluded from the study.

Volunteers will be fasting for 6 hours before sampling to obtain a reproducible alcohol uptake. To avoid dehydration or hypoglycaemia, volunteers will be allowed to drink tea, water or clear fruit juices until 2 hours before sampling.

Blood sampling: from each volunteer two samples of blood will be collected without additives. The first sample (S1) of 14 ml blood will be divided in two halves: 5ml blood for analyzing gut wall integrity without addition of ethanol, the other 5 ml will be analyzed after addition of 5 µl of 96% pure ethanol to obtain a blood concentration of 1‰ ethanol. After the first sample volunteers are randomized to drink either 1 g/kg ethanol in wine (12 gr/100 ml) to obtain a blood alcohol level of 1 ‰ or to drink the same amount in water. The beverages will be consumed in a maximum of 45 minutes. Thirty minutes after the last glass of beverage is consumed, the second sample (S2) of 8 ml blood will be collected. The next 4 samples are taken with one hour intervals (S3, S4, S5 and S6 respectively). The last sample is taken in a second visit at 19:00 the day after. One week after this visit the same protocol will be repeated in which the alcohol and water group will be crossed over.

In each sample I-FABP, L-FABP, LBP, IL-6, ALT, AST, GGT will be measured as well as the alcohol permillage.

Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. Any data collected so far will be destroyed. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

Replacement of individual subjects after withdrawal Replacement of individuals that were withdrawn for whatever reason will take place if necessary. This will be concluded once analysis has been done as this is a pilot study. Replacement will only take place when a subject is not able to complete the protocol.

SAFETY REPORTING In accordance to section 10, subsection 1, of the WMO, the investigator will inform the subjects and the reviewing accredited METC if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal. The study will be suspended pending further review by the accredited METC, except insofar as suspension would jeopardise the subjects' health. The investigator will take care that all subjects are kept informed.

Adverse and serious adverse events Adverse events are defined as any undesirable experience occurring to a subject during the study. All adverse events reported spontaneously by the subject or observed by the investiga¬tor or his staff will be recorded.

A serious adverse event is any untoward medical occurrence or effect that at any dose:

* results in death;
* is life threatening (at the time of the event);
* requires hospitalisation or prolongation of existing inpatients' hospitalisation;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect;
* is a new event of the trial likely to affect the safety of the subjects, such as an unexpected outcome of an adverse reaction, lack of efficacy of an IMP used for the treatment of a life threatening disease, major safety finding from a newly completed animal study, etc.

All SAEs will be reported through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 15 days after the sponsor has first knowledge of the serious adverse reactions.

SAEs that result in death or are life threatening should be reported expedited. The expedited reporting will occur not later than 7 days after the responsible investigator has first knowledge of the adverse reaction. This is for a preliminary report with another 8 days for completion of the report.

Suspected unexpected serious adverse reactions (SUSAR)

Adverse reactions are all untoward and unintended responses to an investigational product related to any dose administered.

Unexpected adverse reactions are adverse reactions, of which the nature, or severity, is not consistent with the applicable product information (e.g. Investigator's Brochure for an unapproved IMP or Summary of Product Characteristics (SPC) for an authorised medicinal product).

The sponsor will report expedited the following SUSARs through the web portal ToetsingOnline to the METC:

* SUSARs that have arisen in the clinical trial that was assessed by the METC;
* SUSARs that have arisen in other clinical trials of the same sponsor and with the same medicinal product, and that could have consequences for the safety of the subjects involved in the clinical trial that was assessed by the METC.

The remaining SUSARs are recorded in an overview list (line-listing) that will be submitted once every half year to the METC. This line-listing provides an overview of all SUSARs from the study medicine, accompanied by a brief report highlighting the main points of concern.

The expedited reporting of SUSARs through the web portal ToetsingOnline is sufficient as notification to the competent authority.

The sponsor will report expedited all SUSARs to the competent authorities in other Member States, according to the requirements of the Member States.

The expedited reporting will occur not later than 15 days after the sponsor has first knowledge of the adverse reactions. For fatal or life threatening cases the term will be maximal 7 days for a preliminary report with another 8 days for completion of the report.

Annual safety report In addition to the expedited reporting of SUSARs, the sponsor will submit, once a year throughout the clinical trial, a safety report to the accredited METC, competent authority, Medicine Evaluation Board and competent authorities of the concerned Member States.

This safety report consists of:

* a list of all suspected (unexpected or expected) serious adverse reactions, along with an aggregated summary table of all reported serious adverse reactions, ordered by organ system, per study;
* a report concerning the safety of the subjects, consisting of a complete safety analysis and an evaluation of the balance between the efficacy and the harmfulness of the medicine under investigation.

Follow-up of adverse events All adverse events will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist.

ETHICAL CONSIDERATIONS Regulation statement The study will be conducted according to the principles of the Declaration of Helsinki (59th WMA General Assembly, Seoul, October 2008 t) and in accordance with the Medical Research Involving Human Subjects Act (WMO) and other guidelines, regulations and Acts

Recruitment and consent All interested persons will receive a folder concerning the study at least two weeks before start of the study. If the volunteer agrees in taking part of the study, the volunteer will be asked to sign the informed consent and take it back to the hospital on the day of the study.

Benefits and risks assessment, group relatedness Subjects consume 1g of alcohol per kg bodyweight. One blood sample of 19 ml followed by 5 samples of 11 ml and one of 8 ml will be drawn between 17.00 hours and 18.00 hours the next day. Observations will take place in two six hour visits and two one hour visits. It is unlikely that subjects will experience any physical or psychological discomfort from the total 82 ml blood sample.

The volunteers will fast for six hours prior to the first blood sample to obtain a reliable blood ethanol concentration. After sampling at 22.00 hours volunteers will be transported homewards by taxi.

Compensation for injury The sponsor/investigator has a liability insurance which is in accordance with article 7, subsection 6 of the WMO.

The sponsor (also) has an insurance which is in accordance with the legal requirements in the Netherlands (Article 7 WMO and the Measure regarding Compulsory Insurance for Clinical Research in Humans of 23th June 2003). This insurance provides cover for damage to research subjects through injury or death caused by the study.

The insurance applies to the damage that becomes apparent during the study or within 4 years after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* male volunteers
* age between 18 and 60 years
* written informed consent

Exclusion Criteria:

* medical history of alcohol abuse
* use of any medication
* medical history of bowel disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The immediate effects of oral alcohol consumption in healthy volunteers on gut wall integrity as measured by I-FABP, LBP and IL-6. | The hours after consumption until 24 hours post-consumption

SECONDARY OUTCOMES:
The immediate effects of oral alcohol consumption in healthy volunteers on the hepatocyte as measured by L-FABP, AST, ALT and GGT. | The hours after consumption until 24 hours post-consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands